CLINICAL TRIAL: NCT02862392
Title: Predictive Progressive Factors of Adolescent Idiopathic Scoliosis
Acronym: SCOLEVOL
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Ecole des hautes études d'ingénieur (HEI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC-P0047
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis
Keywords: Scoliosis; Adolescent; Idiopathic scoliosis; Predictive factors
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of this study is that progressive AIS is characterized by a disorder of orthostatic postural control. The analysis and the treatment of posturographic signal on computerized integrate force plates, coupled to clinical and radiographic examinations, could highlight predictive and reliable factors at the moment of diagnosis. Thus, it could help the clinician in his therapeutic approach, based on the postural control improvement (individualized prescription in kinesitherapy, better adaptation to orthopedic treatments by corset). This method is non-invasive, without side effects, fast and achievable in routine care at the moment of the diagnosis of AIS.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a tridimensional spine deformation affecting 2% of subjects between 10 and 16 years-old being predominant among girls. It is a severe, progressive and multifactorial disease, and a genetic origin is currently admitted.

AIS is progressive (in 3 out of 10 cases) when the scoliosis radiographic frontal angle (Cobb angle) strictly increases by 5° between the diagnosis date and the end of growth. This progression can be severe requiring heavy treatments (corset, surgery) and it can generate adverse effects (spine pain, cardio-respiratory and functional consequences on walking). The lack of reliable criteria to predict the evolution of AIS is a real problem for the therapeutic decision and it can impact the socio-economic cost of the disease.

Several studies show orthostatic postural control anomalies in AIS. The orthostatic postural control is elaborated from the central integration of different sensorial signals (visual, somesthesic and vestibular).

Posturography, on computerized integrate force plates, allows to quantify sensorial components of orthostatic postural control. This technique can confirm the disorders of orthostatic postural control in AIS, but the parameters used can not evaluate with precision the progressive potential.

The posturographic signal analysis could lead to the implementation of therapeutic strategies adapted to progressive risk. Moreover, this method could prevent the progression in major scoliosis, limit the use of radiography, the application of a constraining corset (worn 23 hours a day) and the possibility of heavy surgery (extent arthrodesis).

The hypothesis of this study is that progressive AIS is characterized by a disorder of orthostatic postural control. The analysis and the treatment of posturographic signal on computerized integrate force plates, coupled to clinical and radiographic examinations, could highlight predictive and reliable factors at the moment of diagnosis. Thus, it could help the clinician in his therapeutic approach, based on the postural control improvement (individualized prescription in kinesitherapy, better adaptation to orthopedic treatments by corset). This method is non-invasive, without side effects, fast and achievable in routine care at the moment of the diagnosis of AIS.

ELIGIBILITY:
Inclusion Criteria:

* Female aged from 11 to 14 years
* Patient with AIS, associated with a frontal deviation of spine measured by the radiographic frontal angle of Cobb between 15° and 20°, and a spinal rotation attested by the presence of a gibbosity minimum 5° with Bunnell scoliometer.
* Risser test < 2 (evaluation of the spine bone maturity)
* Patient having front and side views radiographies from spine (huge prints) of less than three months (children have a radiographic check-up from total spine every 6 months on average, no additional print is requested)
* Capable of receiving clear informations
* Giving a written consent for their participation via a consent signed by both parents of the patient (or legal tutor)
* Covered by a healthcare insurance

Exclusion Criteria:

* Patient with secondary scoliosis
* AIS with principal cervico-thoracic curve, according to the Scoliosis Research Society (SRS) classification (this patient category only represents 1% of SIA)
* Primary left thoracic topographic AIS, according to the SRS classification (this category of scoliosis is rare and frequently has a secondary origin: neurologic, polymalformative)
* AIS treated by corrective corset
* Length inequality between inferior members more than 20 mm during clinical examination
* Patient with clinical neurological signs
* Pathological ligamentous laxity
* Known vestibular disease
* BMI > 30
* Refusal to sign an informed consent
* Impossibility to receive clear information

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Female subjects from 11 to 14 years with AIS
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Measure of the evolution of AIS by Recurrence quantification analysis (RQA) | Change from baseline at 24 months
  This parameter allows a posturographic recording of the patient in order to predict the evolution of the disease

SECONDARY OUTCOMES:
Questionnaire to determine presence or absence of family background | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine presence or absence of concomitant illnesses | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine presence or absence of clinical tests of equilibration | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine presence or absence of susceptibility to sensorial conflicts | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine presence or absence of visio-manual laterality | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine type of scoliosis | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine presence or absence of deformed body perception | Change from baseline at 24 months
  For statistical analysis categorical variables may be assigned with numeric indices
Questionnaire to determine date of first periods | Change from baseline at 24 months
  Questionnaire to determine date of first periods
Quantification of body mass index | Change from baseline at 24 months
  Quantification of body mass index
Questionnaire to determine presence or absence of socio-demographic variables | at baseline
  For statistical analysis categorical variables may be assigned with numeric indices
Fukuda stepping test in order to evaluate the vestibular sensory input | Change from baseline at 24 months
  The purpose of the Fukuda Stepping Test (FST) is to measure asymmetrical vestibulospinal reflex tone resulting from labyrinthine dysfunction
Pearson correlation coefficient to determine the correlation between posturographic and radiographic parameters | Change from baseline at 24 months
  Pearson correlation coefficient to determine the correlation between posturographic and radiographic parameters
Score of the motion Sickness Susceptibility Questionnaire | Change from baseline at 24 months
  Score of the motion Sickness Susceptibility Questionnaire
Trunk Appearance Perception Scale | Change from baseline at 24 months
  Evaluation of self appearance or image

CONTACTS AND LOCATIONS:
Overall Officials: Catanzariti Jean-François, MD, Principal Investigator — Lille Catholic University; Olivier Agnani, Study Chair — Lille Catholic University
Locations (4):
- France (4):
  - Fondation Hopale, Berck, Hauts-de-France
  - Centre de MPR pour enfants de Bois Larris, Lamorlaye, Hauts-de-France
  - SSR pédiatrique Marc Sautelet, Villeneuve-d'Ascq, Hauts-de-France
  - CHU d'Amiens, Amiens, Picardie

IPD SHARING:
Plan to Share IPD: No